CLINICAL TRIAL: NCT02644200
Title: Gelatin Tannate as Treatment for Acute Childhood Gastroenteritis: a Prospective, Randomized, Single-blind Controlled Clinical Trial
Brief Title: Gelatin Tannate as Treatment for Acute Childhood Gastroenteritis
Acronym: GT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Marina Aloi, MD, PhD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2015
Record Dates: First submitted 2015-12-16; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Acute Gastroenteritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ORS (No Intervention): Controls treated with oral rehydration solution (standard therapy)
- ORS+GT (Active Comparator): Group treated with oral rehydration solution plus gelatin tannate
  Interventions: Device: Gelatin tannate

INTERVENTIONS:
Device: Gelatin tannate
  Other Names: Gelenterum
  Arms: ORS+GT

SUMMARY:
Oral rehydration therapy is the only treatment recommended by the World Health Organization in acute diarrhea in children. The aim of this study was to compare the efficacy and safety of a therapy with gelatin tannate plus oral rehydration versus oral rehydration alone in children with acute gastroenteritis.

This is a single-blind, prospective, randomized and parallel study performed in two Pediatric Services of tertiary referral hospitals. Patients, ages 3 to 36 months with acute gastroenteritis randomized to receive an oral rehydration solution (OR), or an oral rehydration solution plus gelatin tannate (OR+G). The primary outcomes evaluated were: the number of bowel movements after 48 and 72 hours after initiating treatments. Secondary outcomes were: duration of diarrhea (days), stool characteristics and adverse events. Other clinical variables, as weight, fever, vomiting, appetite and the acceptability of the two treatments were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sex, aged 3 months to 5 years of age
* Clinical diagnosis of acute gastroenteritis, as defined by having at least 3 loose stools within the previous 24 hours and/or a change in stool consistency to loose or liquid according to Bristol Stool Form Scale for Children (m-BSFS-C) lasting for no longer than 3 days.

Exclusion Criteria:

* patients with gastroenteritis lasting more than 5 days
* patients with chronic gastrointestinal conditions
* patients receiving other antidiarrheal drugs within 2 weeks prior to enrollment (i.e. antibiotics, probiotics, salicylates, loperamide, racecadotril, disomectite)

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of stools | 48 hours
  difference in the number of stools after treatment initiation in the 2 arms

SECONDARY OUTCOMES:
Duration of diarrhea after treatment initiation in the 2 arms | 48 hours, 72 hours
  The duration of diarrhea was defined as the time in hours from enrolment to the last abnormal (loose or liquid) stool. Last abnormal stool was defined when the child passed to normal stool or no stool for next 24 hours
Time to normalization of stool consistency | 48 hours, 72 hours
  Stool consistency was evaluated on a modified Bristol Stool Form Scale for Children (m-BSFS-C) and defined as: 1: separate hard lumps, like nuts; 2: Sausage-shaped but lumpy; 3: like a sausage or snake, smooth and soft; 4: fluffy pieces with ragged edges, a mushy stool; 5: watery, no solid pieces
Number of visits to the emergency room | 7 days
  need for additional visits during the 7 days of treatment in the 2 arms
Growth | 7 days
  growth parameters in the 2 arms
Adverse events treatment related | 7 days
  Number of participants with drug-related adverse events in the 2 arms

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Sapienza University of Rome, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mennini M, Tolone C, Frassanito A, Midulla F, Cucchiara S, Aloi M. Gelatin Tannate for Acute Childhood Gastroenteritis: A Randomized, Single-Blind Controlled Trial. Paediatr Drugs. 2017 Apr;19(2):131-137. doi: 10.1007/s40272-016-0207-z. PMID 28000174